CLINICAL TRIAL: NCT04182880
Title: Phase 2a, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety and Pharmacokinetic Profile of CPL-01 in the Management of Acute Postoperative Pain After Mini-abdominoplasty Surgery
Brief Title: Evaluate the Safety and Pharmacokinetic Profile of CPL-01 in the Management of Acute Postoperative Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cali Pharmaceuticals LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CPL-01_AB_001
Record Dates: First submitted 2019-11-26; First posted 2019-12-02 (Actual); Results first posted 2022-09-21 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-08

CONDITIONS: Abdominoplasty

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- CPL-01 (Experimental): CPL-01
  Interventions: Drug: CPL-01

INTERVENTIONS:
Drug: CPL-01 — CPL-01 will be administered
  Arms: CPL-01
Drug: Placebo — Placebo will be administered
  Arms: Placebo

SUMMARY:
Evaluate the Safety and Pharmacokinetic Profile of CPL-01 in patients after mini-abdominoplasty

DETAILED DESCRIPTION:
This is a randomized, double-blind, study to evaluate the safety, PK profile of CPL-01 for the management of postoperative pain after mini-abdominoplasty surgery.

ELIGIBILITY:
Inclusion Criteria:

* Subject provides signed, written informed consent before participation in the study.
* Subject is aged ≥18 and ≤70 years at the time of informed consent and is male or female.
* Subject is scheduled to undergo elective mini-abdominoplasty surgery under general anesthesia without collateral procedures.
* Female subjects are eligible only if all the following apply:

  1. Not pregnant
  2. Not breastfeeding
  3. Not planning to become pregnant during participation in the study
  4. Committed to the use of an acceptable form of birth control for the duration of the study until at least 30 days after administration of IP.
* Male subjects must commit to the use of a reliable method of birth control for the duration of the study until at least 30 days after administration of IP or be surgically sterile (biologically or surgically).
* Subject is free of any physical, mental, or medical conditions which, in the opinion of the investigator, make mini-abdominoplasty or study participation inadvisable.

Exclusion Criteria:

* Subject has known, suspected, or reported history of alcohol or drug abuse or dependence within the previous 2 years as assessed by the investigator
* Subject has impaired liver function (e.g., aspartate aminotransferase/alanine aminotransferase greater than 3 times the upper limit of the reference range, bilirubin greater than 1.5 times the upper limit of the reference range unless due to Gilbert's syndrome, active hepatic disease, evidence of clinically significant liver disease, or other condition such as alcoholism, cirrhosis, or hepatitis, etc.) that suggests the potential for an increased susceptibility to hepatic toxicity with IP exposure.
* Subject has clinically significant renal abnormalities (creatinine ≥1.5 × upper limit of normal).
* Subject has hemoglobin A1c ≥7.0%.
* Subject has participated in another clinical study and/or received an IP (marketed or premarket) within 30 days before surgery.
* Subject has a history of, or positive test results for, human immunodeficiency virus, hepatitis B surface antigen, or hepatitis C virus antibody at Screening.
* Subject with an upper respiratory infection/cough in the 14 days before surgery.
* Subjects with a history of significant postoperative nausea and vomiting.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erol Onel, MD, Study Chair — Cali Biosciences
Locations (1):
- Chesapeake Research Group, Pasadena, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | CPL-01
Started | 5 | 15
Completed | 4 | 15
Not Completed | 1 | 0
Not completed — Pregnancy | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | CPL-01 | Total
Number analyzed (Participants) | 5 | 15 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 15 | 20
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 15 | 20
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 15 | 20
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 13 | 17
  White | 0 | 2 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean (Peak) Plasma Concentration (Cmax)
Description: Mean Cmax of 573 ng/mL and occurred at approximately 13 hours. Timepoints tested included before study drug administration and 15, 30, and 45 minutes and 1, 2, 4, 6, 8, 10, 12, 18, 24, 30, 36, 48, 60, 72, 96, and 120 hours after administration.
Time Frame: Baseline through 120 hours after start of study drug administration
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Placebo | CPL-01
Number analyzed (Participants) | 5 | 15
ng/mL | 0 (0) | 573 (258)

ADVERSE EVENTS:
Time Frame: 28 Days
Arm/Group | Placebo | CPL-01
All-Cause Mortality (participants affected / at risk) | 4/5 | 11/15
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/15
Other Adverse Events (participants affected / at risk) | 4/5 | 11/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=5) | CPL-01 (N=15)
Nausea (Gastrointestinal disorders) | 1 (1) | 3 (3)
Constipation (Gastrointestinal disorders) | 1 (1) | 4 (4)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Feeling Hot (General disorders) | 1 (1) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 2 (2) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Bacterial Vaginosis (Infections and infestations) | 1 (1) | 0 (0)
Incision Site Rash (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-11-25): https://cdn.clinicaltrials.gov/large-docs/80/NCT04182880/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-07): https://cdn.clinicaltrials.gov/large-docs/80/NCT04182880/SAP_001.pdf